CLINICAL TRIAL: NCT02387736
Title: Dialectical Behaviour Therapy for Chronically Self-harming Individuals With BPD: Evaluating the Clinical and Cost Effectiveness of a 6-month Treatment
Brief Title: DBT for Chronically Self-harming Individuals With BPD: Evaluating the Clinical & Cost Effectiveness of a 6 mo. Treatment
Acronym: FASTER-DBT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Simon Fraser University (Other)
Responsible Party: Principal Investigator, Shelley McMain, Head, Borderline Personality Disorder Clinic, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 026/2014
Record Dates: First submitted 2015-02-20; First posted 2015-03-13 (Estimated); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Borderline Personality Disorder
Keywords: BPD; DBT; Dialectical Behaviour Therapy; Borderline Personality Disorder; Suicide; Non-suicidal self injury; NSSI; Randomized Control trials; treatment
MeSH Terms: conditions — Borderline Personality Disorder; Suicide; Self-Injurious Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dialectical Behaviour Therapy-6 months (Experimental): 6 months of standard dialectical behaviour therapy treatment.
  Interventions: Behavioral: Dialectical Behaviour Therapy-6 months
- Dialectical Behaviour Therapy-12 months (Active Comparator): 12 months of standard dialectical behaviour therapy treatment
  Interventions: Behavioral: Dialectical Behaviour Therapy-12 months

INTERVENTIONS:
Behavioral: Dialectical Behaviour Therapy-6 months — Modification of behaviours achieved with reframing thoughts and impulses
  Other Names: DBT-6
  Arms: Dialectical Behaviour Therapy-6 months
Behavioral: Dialectical Behaviour Therapy-12 months — Modification of behaviours achieved with reframing thoughts and impulses
  Other Names: DBT-12
  Arms: Dialectical Behaviour Therapy-12 months

SUMMARY:
Standard one-year dialectical behaviour therapy (DBT), which has four components, is an effective treatment for people with borderline personality disorder. However, such DBT programs are in short supply and costly, resulting in long wait lists. In practice, DBT is often reduced in length or intensity. This study will determine whether shorter DBT treatment is clinically effective and cost-effective. In total, 240 self-harming BPD patients will be randomly assigned to receive either 1 year or 6 months of DBT, with follow-up lasting two years. Rates of suicidal and self-harm behaviours, use of health care and general psychological functioning will be examined.

DETAILED DESCRIPTION:
Borderline personality disorder (BPD) is a serious and debilitating psychiatric condition characterized by instability in relationships, emotions, identity, and behaviour. Affecting 2-6% of the general population, BPD is associated with high rates of self-harm (both suicide attempts and non-suicidal self-injury), mortality by suicide, and consequent heavy use of public health resources, making it one of the most expensive psychiatric disorders to treat. Psychotherapy is recognized as the first-line treatment for BPD, of which dialectical behaviour therapy (DBT) has demonstrated the strongest empirical support. Although DBT is efficacious for self-harming individuals with BPD, and increasingly available over the past 10 years, demand for DBT exceeds existing resources.

Within the current climate of rising health care costs and limited resources, the length (12 month) and intensive nature (entailing multiple treatment components) of standard DBT are major barriers to its adoption. Subsequently, most DBT programs have lengthy wait lists. Inadequate accessibility of treatment is not specific to Canada; it is a global problem. In clinical practice, DBT is often abbreviated, or clinicians deliver only the components that they believe are most appropriate, despite an evidence base almost entirely consisting of studies of 1 year of DBT. There are no data on the optimal length of treatment.

Therefore, the primary aim of this proposal is to examine the efficacy of an abbreviated course of DBT (including all components of treatment) compared to the evidence-supported 12 months of DBT. Our principal question is: How do the clinical outcomes of 6 months of DBT (DBT-6) compare with the standard 12 months (DBT-12) for the treatment of chronically self-harming individuals with BPD? Assessments will be conducted at pretreatment and at 3-month intervals until 24 months (i.e., 3, 6, 9, 12, 15, 18, 21, and 24 months).

Hypotheses: (1) Patients in the DBT-6 arm will show reductions in the frequency of self-harm across the treatment phase and one-year post treatment follow-up phase no worse than those measured with patients in the DBT-12 arm. (2) Patients who present with high rates of self-harm and impulsive behaviours will have reductions in the frequency of self-harm behaviours that are no worse than those in the DBT-6 arm and the DBT-12 arm, over the course of both the treatment phase and the 1-year post treatment follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for Borderline Personality Disorder.
* Has had at least 2 self-harm episodes (either suicidal or non-suicidal) in the past 5 years, including at least 1 in the past 8 weeks.
* Proficient in English
* Provides informed consent to participate in the study.
* Absence of 8 or more standard weeks of DBT in the past year (individual and group therapy components).
* has had either Ontario Health Insurance Plan (OHIP) coverage or BC Medical Services Plan (MSP) health insurance for 1 year or more
* Absence of a pending criminal court case or charges.
* Has been a resident of Ontario or British Columbia for all of the past 12 months, at least.
* Lives in the Greater Toronto Area/Greater Vancouver Area

Exclusion Criteria:

* Meets the DSM-IV criteria for bipolar disorder I, dementia, or a psychotic disorder other than psychotic disorder NOS
* IQ less than 70
* Chronic or serious physical health problem requiring hospitalization within the next year (e.g., cancer)
* Plans to move to a province other than Ontario or BC in the next 2 years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Change in frequency of self-harm (suicidal and non-suicidal) behaviours over time as measured by the Suicide Attempt Self-Injury Interview (SASII) | Administered pre-treatment and every three months until 24 months
  Records details regarding the frequency, topography, intent, medical severity, social context, precipitating and concurrent events, and outcomes of each self-harm (suicidal and non-suicidal) behavior during a three-month target time period.

SECONDARY OUTCOMES:
Changes in health care use as measured by the Treatment History Interview-2 (THI-2) | Administered pre-treatment and every three months until 24 months
  Records participants use of other treatment resources, e.g. number of Hospitalizations, Emergency Room Visits, Medications, Psychosocial Treatments
Change in general functioning as measured by the Euroqol-5D | At pre-treatment and every three months until 24 months
  Assesses health related quality of life
Change in BPD symptoms as measured by the Borderline Symptom List-23 (BSL-23) | At pre-treatment and every three months over 24 months
  Assesses presence of specific BPD symptoms
Change in general psychopathology and symptoms, as measures by the Symptom Checklist 90 Revised (SCL-90R) | At pre-treatment and every three months over 24 months
  Assesses general symptom distress
Change in anger as measured by the State-Trait Anger Expression Inventory-2 (STAXI-2) | At pre-treatment and every three months over 24 months
  Assesses a subject's experience and expression of anger
Change in depression as measured by the Beck Depression Inventory-II (BDI-II) | At pre-treatment and every three months over 24 months
  Assesses symptoms of depression
Changes to interpersonal functioning as measured by the Inventory of Interpersonal Problems-64 (IIP-64) | At pre-treatment and every three months over 24 months
  Assesses dysfunctional patterns in interpersonal interactions
Changes in the use of DBT coping skills, as measured by the Dialectical Behaviour Therapy Ways of Coping Checklist (DBT-WCCL) | At pre-treatment and every three months over 24 months
  Assesses the use of DBT skills

CONTACTS AND LOCATIONS:
Overall Officials: Shelley McMain, Ph.D, Principal Investigator — The Centre for Addiction and Mental Health
Locations (2):
- Canada (2):
  - Simon Fraser University, Burnaby, British Columbia
  - Center for Addiction and Mental Health, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Psychiatric Association. Diagnostic and Statistical Manual of Mental Disorders 2013; 5 ed. Washington, DC: American Psychiatric Association Press.
- [Background] Grant BF, Chou SP, Goldstein RB, Huang B, Stinson FS, Saha TD, Smith SM, Dawson DA, Pulay AJ, Pickering RP, Ruan WJ. Prevalence, correlates, disability, and comorbidity of DSM-IV borderline personality disorder: results from the Wave 2 National Epidemiologic Survey on Alcohol and Related Conditions. J Clin Psychiatry. 2008 Apr;69(4):533-45. doi: 10.4088/jcp.v69n0404. PMID 18426259
- [Background] Soeteman DI, Hakkaart-van Roijen L, Verheul R, Busschbach JJ. The economic burden of personality disorders in mental health care. J Clin Psychiatry. 2008 Feb;69(2):259-65. doi: 10.4088/jcp.v69n0212. PMID 18363454
- [Background] Bateman AW. Treating borderline personality disorder in clinical practice. Am J Psychiatry. 2012 Jun;169(6):560-3. doi: 10.1176/appi.ajp.2012.12030341. No abstract available. PMID 22684591
- [Background] Skodol AE, Gunderson JG, Pfohl B, Widiger TA, Livesley WJ, Siever LJ. The borderline diagnosis I: psychopathology, comorbidity, and personality structure. Biol Psychiatry. 2002 Jun 15;51(12):936-50. doi: 10.1016/s0006-3223(02)01324-0. PMID 12062877
- [Background] Skodol AE, Siever LJ, Livesley WJ, Gunderson JG, Pfohl B, Widiger TA. The borderline diagnosis II: biology, genetics, and clinical course. Biol Psychiatry. 2002 Jun 15;51(12):951-63. doi: 10.1016/s0006-3223(02)01325-2. PMID 12062878
- [Background] Black DW, Blum N, Pfohl B, Hale N. Suicidal behavior in borderline personality disorder: prevalence, risk factors, prediction, and prevention. J Pers Disord. 2004 Jun;18(3):226-39. doi: 10.1521/pedi.18.3.226.35445. PMID 15237043
- [Background] Comtois, K. A., Elwood, L., Holdcraft, L. C., Smith, W. R., Simpson, T. L. Effectiveness of dialectical behaviour therapy in a community mental health centre. Cognitive And Behavioral Practice 2007; 14(4):406-14.
- [Background] Bateman A, Fonagy P. Health service utilization costs for borderline personality disorder patients treated with psychoanalytically oriented partial hospitalization versus general psychiatric care. Am J Psychiatry. 2003 Jan;160(1):169-71. doi: 10.1176/appi.ajp.160.1.169. PMID 12505818
- [Background] Zanarini MC, Frankenburg FR, Hennen J, Silk KR. Mental health service utilization by borderline personality disorder patients and Axis II comparison subjects followed prospectively for 6 years. J Clin Psychiatry. 2004 Jan;65(1):28-36. doi: 10.4088/jcp.v65n0105. PMID 14744165
- [Background] McMain SF, Links PS, Gnam WH, Guimond T, Cardish RJ, Korman L, Streiner DL. A randomized trial of dialectical behavior therapy versus general psychiatric management for borderline personality disorder. Am J Psychiatry. 2009 Dec;166(12):1365-74. doi: 10.1176/appi.ajp.2009.09010039. Epub 2009 Sep 15. PMID 19755574
- [Background] Linehan MM, Comtois KA, Murray AM, Brown MZ, Gallop RJ, Heard HL, Korslund KE, Tutek DA, Reynolds SK, Lindenboim N. Two-year randomized controlled trial and follow-up of dialectical behavior therapy vs therapy by experts for suicidal behaviors and borderline personality disorder. Arch Gen Psychiatry. 2006 Jul;63(7):757-66. doi: 10.1001/archpsyc.63.7.757. PMID 16818865
- [Background] McMain SF, Guimond T, Streiner DL, Cardish RJ, Links PS. Dialectical behavior therapy compared with general psychiatric management for borderline personality disorder: clinical outcomes and functioning over a 2-year follow-up. Am J Psychiatry. 2012 Jun;169(6):650-61. doi: 10.1176/appi.ajp.2012.11091416. PMID 22581157
- [Background] Linehan, M.M. Cognitive Behavioural Treatment of Borderline Personality Disorder. New York: Guilford Press; 1993.
- [Derived] Christensen KE, McMain S, Chapman A, Kuo JR. An examination of the role of PTSD and childhood trauma on treatment outcomes for individuals with borderline personality disorder in dialectical behavior therapy. Borderline Personal Disord Emot Dysregul. 2025 Nov 12;12(1):47. doi: 10.1186/s40479-025-00322-2. PMID 41225564
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793
- [Derived] McMain SF, Chapman AL, Kuo JR, Guimond T, Streiner DL, Dixon-Gordon KL, Isaranuwatchai W, Hoch JS. The effectiveness of 6 versus 12-months of dialectical behaviour therapy for borderline personality disorder: the feasibility of a shorter treatment and evaluating responses (FASTER) trial protocol. BMC Psychiatry. 2018 Jul 17;18(1):230. doi: 10.1186/s12888-018-1802-z. PMID 30016935
- See also: The Centre for Addiction and Mental Health (CAMH) is the leading mental health and addictions research facility in Canada, and one of the largest in the world. — http://www.camh.ca/en/research